CLINICAL TRIAL: NCT06130488
Title: Implementation at Scale and Evaluation of KMC (Kangaroo Mother Care)
Brief Title: Implementation at Scale and Evaluation of KMC
Acronym: KMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Distinguish Professor, Aga Khan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-6444-19970
Record Dates: First submitted 2022-11-28; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Newborn Morbidity
Keywords: Low birth weight; Kangaroo Mother Care; Newborn care

STUDY DESIGN:
Intervention Model Description: Quasi experimental study model with pre and post intervention evaluation,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KMC implementation (Experimental): KMC phases implemented as per the protocol
  Interventions: Behavioral: KMC

INTERVENTIONS:
Behavioral: KMC — KMC implementation as per protocol

SUMMARY:
The goal of this quasi-experimental study design is to look at feasibility and document the process and challenges of implementing KMC at scale in district Sanghar (Sindh) and Lasbella (Balochistan)

. The main question it aims to answer are:

* Does the KMC is feasible to be implemented in rural areas?
* What is the process and challenges in implementing KMC in rural areas?
* Pregnancy surveillance is going in the secondary level care hospitals and in its catchment population. Recruitment of babies is carried who are low birth weight (less than 2000grams).
* Mothers taught to administer KMC by physician and nursing /LHV staff in the facility within first 6 hours after delivery and continue till the mother and baby are discharged by trained facility KMC management team.
* After training and administration of KMC at facility for 72 hours, the mother and baby pair discharged and followed up at home by the team including project-based data collector and respective LHWs.
* KMC Champions are in development for community mobilization and conducting sessions at village level.
* We will compare pre and post intervention change in practices at facility level and at individual level of household and assess the KMC coverage.

DETAILED DESCRIPTION:
KMC Implementation

Pre KMC-Implementation phase (Community) Birth weight of all newborns in selected facilities and home will be captured by trained lady health workers (LHW)/community health workers (CHW) with digital scales. LHW/CHW will refer all 2000 g or less newborns to facilities for KMC. LHWs will create community awareness and engagement to support and accept referral of newborns for KMC through Village Health committee members (VHC) and by approaching existing women support groups formed by LHWs during phase 1 of the project.

KMC Implementing Facilities

Training of Staff A total of 40 facility-based health care providers and 400 community-based workers including LHWs/ LHVs in Sanghar and Lasbela will receive a three-day training session on KMC & Essential newborn care followed by a one-day training on DHIS data record keeping.

KMC Facilities Preparation: Sustainable Provision of KMC and Essential Commodities/supplies Spaces already present within the selected facilities will be identified to serve as KMC rooms (curtained/ partitioned areas, toilets), so mothers can stay with their babies. Facilities will contain essential equipment for maternal and newborn care such as ambu bags, weighing scales for newborns, KMC packs, infant heaters, oxygen supply systems and pulse oximeters.

Methodology

Study Design:

We have carried out formative research to identify barriers and design a model to deliver KMC across the facility-community continuum. A quasi-experimental study design will be adopted. District Health Information System (DHIS) data and service data on maternal and newborn mortality and morbidity outcomes will be collected from health facilities. A pre and post design will be undertaken to look at feasibility and document the process and challenges of implementing this at scale.

Study population The study population are babies of birth weight less than 2000g delivered at hospital or in community in the catchment area of 2 district in Sindh and Balochistan.

Study settings and location:

This model will be implemented in the facilities and their catchment communities of district Sanghar and district Lasbela from July 2021 for 24 months. Four tehsils will be selected from each district, health facilities accompanying in these tehsils are already identified along with their catchment population to implement community arm of KMC. The facilities that will implement KMC include DHQs, THQs and RHCs from public sector and private sector facilities. And these facilities have been selected based on the availability of MNCH services and logistics. These facilities are level two hospitals (DHQs & THQs) and MNCH centers (RHCs) equipped with essential equipment's, supplies, drugs, basic laboratory test, immediate referral and human resources. The monthly outpatient turnover of the maternal patients in each of these hospitals on average 80 - 120 deliveries for DHQs and THQs takes place each month.

Study Activities

Base line Survey:

The UeN midline survey will be used as baseline for this research and end-line surveys will be conducted in 2023. The community KMC indicators will be; prevalence of low birth weight babies, neonatal mortality, KMC practices, skin-skin contact, breast feeding practices, immediate and essential newborn care practices, especial care of low birth weight babies provided by families and care seeking behavior for newborns.

Pregnancy surveillance:

Pregnancy surveillance will be instituted through LHWs for detection of new pregnancies as a continuous monthly activity throughout the study period. Families will be encouraged for facility-based delivery and KMC will be administered to all Low-birth-weight babies (<2000gms) delivered in the facility. The Pregnancy surveillance data will be validated by data collectors during their monthly visit for Birth notification. Identified pregnancies will be followed up by data collectors who will monitor sessions on KMC at household level to orient pregnant mother and their families on KMC benefits, conducted by respective LHW. This will be an antenatal sensitization activity. As soon as a home birth is notified, district-based project staff will ensure LHW will visit the household within 72 hours of birth. The screening will be carried out and babies with birth weight of 2000 gram or less will be referred to KMC facility. After discharge from facility, the LHW will visit the household on (days 7, 14, 21, and 28) and district team validate these visits to assess the mother and baby and support kangaroo mother care practice.

Enrollment and KMC administration at Facility:

Low birth weight babies (<2000gms) delivered in facility will be enrolled at birth if they fulfill eligibility criteria and following consent. KMC will be administered to all enrolled babies. Mothers will be taught to administer KMC by physician and nursing /LHV staff in the facility within first 6 hours after delivery and will continue till the mother and baby are discharged by trained facility KMC management team.

Continuation of KMC administration at Community:

After training and administration of KMC at facility for 72 hours, the mother and baby pair will be discharged and followed up at home by the team including project-based data collector and respective LHWs. Team will conduct follow up visits daily for the first week, then weekly basis for 6 weeks, then quarterly till 2 years of age to capture process indicators. Data collectors will visit all households in the tehsils on the scheduled basis to ensure support for providing KMC and reinforcement. For women who deliver low birth weight babies at home, window period for enrolment will be 72 hours. KMC will be taught to them at home by LHWs and validated by project-based staff. Their responsibility will be to support mothers in practicing KMC. Community based Kangaroo Mother Care (cKMC) will be administered by LHWs only to enrolled babies discharged from facilities and those born at home belonging to the catchment population of already identified KMC facilities.

Community Mobilization (KMC Champions):

KMC Champions will be developed for community mobilization and conducting sessions at village level. LHW / CHW with the support of village health committee and support groups will also conduct one-to-one and group sessions with pregnant women, mothers and mothers-in-law on essential newborn care and KMC practices. The sessions will be conducted at regular intervals which validated and monitored by project-based district managers. LHW/CHW will also encourage recruitment of volunteers to function as KMC champions. The local community members serving as KMC champions will also serve as catalyst for mobilization. The mobilization staff will also identify and encourage co-champions (a stream of volunteers from the community) who will be mentored by KMC champions. This group of local community members will serve to disseminate messages on KMC practices and to facilitate its uptake in the community.

Data Collection A data collection team consisting of 2 members will be instituted for each implementing tehsils. Their responsibility will be to collect data on the process indicators weekly for the first 6 weeks and then quarterly till 2 years.

Impact Assessments A midline assessment will be done at all facilities and their catchment populations in all tehsils after one year of intervention. This midline assessment will serve to provide us with outcomes and evaluation of the intervention. Results of midline will identify areas of improvement and re-modeling if needed. A final assessment will be carried out after the completion of (Facility KMC plus cKMC) intervention in all tehsils. Through this design we will compare pre and post intervention change in practices at facility level and at individual level of household. End line assessment will be carried out to estimate increase in effective coverage of KMC among newborns having birth weight of 2000grams or less.

Training of Facility and Community Providers This implementation project will be guided by the experience of our Dadu-KMC project, and we will adopt the contextual insights and the information, education and counselling material used in the project for parents and families to create awareness and to explain the benefits of KMC for survival & wellbeing of low-birth-weight newborns.

Facility Based KMC Facility based Kangaroo Mother Care (KMC) will be practiced at health facilities, where newborns are delivered or referred. The frontlines workers are health professional involved in newborn care will be trained such as physicians, nurses, midwives, technicians and obstetricians at facility level. The training will be conducted over 3-4 days. The content will include the theoretical knowledge as well as teaching the complete set of skills. Information, Education and Communication material will be used for implementing KMC at the facility. The IEC material will include messages in the pictorial form on KMC positioning, nutrition (breast feeding, feeding expressed breast milk or feeding through nasogastric tube), criteria for discharge, monitoring and assessment during KMC, recognition of danger sings, referral and follow-up. Recording tools will be adapted and developed to record the observations when implementing KMC at the facility level. The IEC material is comprised of flip charts, wall mounts and a self-explanatory video on steps of KMC, its benefits.

Community Based KMC Community KMC will be practiced at the household levels where newborns are cared by mother, father and family members. Health Providers from the community such as LHWs will visit households and assess babies according to the scheduled follow-up visits. At community level mother, spouse, family members, community leaders, LHVs, LHWs, CHWs, and TBAs, which will be trained first for community KMC.

Experts from AKU will serve as trainers for KMC and essential newborn care. Educational material such as information, pictorial booklet, flip charts and video films on KMC in local language will be made available for the mothers, families, facility providers, LHWs and study staff. These trainings will be conducted at the field site, through KMC videos and flip charts. The training routine will consist of 2-day classroom and 2 day real life field scenario for facility providers. Similarly, the LHW's of the selected facility catchment area will also be trained to pregnancy surveillance, case referral, notification and follow-ups and will also be trained to deliver information, education and support for the KMC practices at the household level in 2 days training workshop by respective facility providers.

ELIGIBILITY:
Inclusion Criteria:

• Baby weighing between ≥1200 to <2000grams

Exclusion Criteria:

* Well small baby; less than 1200 grams
* Baby more than 2000g
* Danger signs such as
* Severe infections
* Apnea
* Congenital malformation

Ages: 30 Minutes to 42 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2500 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Number of infants having birth weight of 2000 grams received Kangaroo Mother Care (KMC) | Through study completion, average 2 years
  Low Birth weight (<2000grams) infants enrolled and received at the implementation sites (secondary level care hospitals and their catchment population) in two districts

SECONDARY OUTCOMES:
Increase in exposure to KMC priming interactions in the antenatal period | Through study completion, average 2 years
  (i) Proportion of identified pregnant women who received KMC information in the antenatal period from LHWs (either at home visits or during planned community interactions, (ii) Proportion of identified pregnant women who received KMC information during ANC visits at health facilities
Proportion of the health facilities providing KMC services | Through study completion, average 2 years
  Having dedicated KMC space with appropriate staffing, supplies and guidelines
Number of infants received early Initiation and Exclusive breast feeding | Through study completion, average 2 years
  Breastfeeding within1 hour is early initiation of breastfeeding. Exclusive Breastfeeding is the continue breast fed till 6 months of newborns without giving any thing else.

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar Bhutta, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
All identified information of the study participants will be kept confidential. It may only be accessed by the principal investigators or supervisors.